CLINICAL TRIAL: NCT05850221
Title: Anaerobic Exercise as a Modulator of Microbial Composition and Mental Acuity in Sedentary Men
Brief Title: Anaerobic Exercise and Mental Acuity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00017316
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Depression; LPS; Mood
MeSH Terms: conditions — Depression | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: randomized controlled trial (waitlist control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weight training (Experimental): A prescribed 8-week training protocol
  Interventions: Other: weight training
- no prescribed weight training (No Intervention): no prescribed weight training

INTERVENTIONS:
Other: weight training — weight training
  Arms: weight training

SUMMARY:
This is a randomized controlled trial to examine the effect of anaerobic activity (e.g., weight training) on gut microbiome metabolism and neurological health in healthy sedentary men.

DETAILED DESCRIPTION:
The human gut microbiome, which houses over 2,000 distinct bacterial species, has recently been characterized as a highly influential force on the health and longevity of its host. By way of several distinct pathways comprising the "microbiome-gut-brain axis", this diverse population is known to communicate with the human brain in a bidirectional manner and is implicated in the pathophysiology of several metabolic and psychological disease states. The ability to support a healthy, diverse microbiome through modifiable behavioral interventions - such as diet and exercise - is a topic of growing interest. Most of the evidence pertaining to the relationship between physical activity and the gut-brain axis at this time, however, investigates the influence of aerobic exercise providing limited insight to how other modalities of physical activity may differ. Specifically, this study will examine the impact of an 8-week weight training protocol on gut microbiome metabolism and neurological health in healthy sedentary men. Participants will be randomly assigned to the intervention group or the waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

* free of any existing medical diagnoses
* willing and able to participate in moderate to vigorous exercise as determined by the ACSM Health/Fitness Facility Preparticipation Screening Questionnaire
* sedentary (defined as a score <14 on the Godin-Shepard Leisure Time Physical Activity Questionnaire (GSLTQ))
* equipped with access to a complete gym

Exclusion Criteria:

* antibiotic use within the past six months
* prebiotic, probiotic, or high-dose antioxidant supplementation within the past 6 months
* smoker (cigarettes and/or marijuana)
* regular laxative use
* blood pressure >129/80 at baseline

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
gut barrier integrity | change from baseline at week 8
  serum LPS binding protein

SECONDARY OUTCOMES:
mood state | change from baseline at week 8
  Depression score on Center for Epidemiological Studies-Depression (CES-D) questionnaire.
  Scores range from 0-60, with scores >15 indicating an elevated risk of depression and scores >30 indicating elevated symptoms of depression that may influence the health of the individual

OTHER OUTCOMES:
anaerobic capacity | change from baseline at week 8
  wingate test

CONTACTS AND LOCATIONS:
Locations (1):
- 850 PBC, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No